CLINICAL TRIAL: NCT04156516
Title: Longitudinal Effects of a Sexual Health Intervention: HEART
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic interfered with school-based data collection
Sponsor: North Carolina State University (Other)
Responsible Party: Principal Investigator, Laura Widman, Associate Professor of Psychology, North Carolina State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 55597
Record Dates: First submitted 2019-11-02; First posted 2019-11-07 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: STD; Adolescent Behavior
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEART (Experimental): sexual health intervention that focuses on communication skills
  Interventions: Behavioral: HEART
- HealthyMinds (Active Comparator): Attention-matched control: Growth mindset intervention
  Interventions: Behavioral: HealthyMinds

INTERVENTIONS:
Behavioral: HEART — sexual health intervention
  Arms: HEART
Behavioral: HealthyMinds — Growth mindsets of personality and mental health
  Arms: HealthyMinds

SUMMARY:
Randomized Controlled Trial to evaluate the eHealth program, HEART (Health Education and Relationship Training).

DETAILED DESCRIPTION:
Randomized Controlled Trial to evaluate the eHealth program, HEART (Health Education and Relationship Training). Data collection will occur at pretest, posttest, 12m (primary endpoint) and 18m (to look at stability of effects over time).

ELIGIBILITY:
Inclusion Criteria:

* Current high school student
* Able to read English

Exclusion Criteria:

* Not able to read English

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Condom use at last sex | 12 months
  Percentage of participants who used condoms at last sexual intercourse in the treatment group compared to the control group
Sexual intercourse within the past 12 months | 12 months
  Percentage of participants who had sexual intercourse in the past 12 months in the treatment group compared to the control group

SECONDARY OUTCOMES:
HIV/STD Knowledge | 12 months
  9-item HIV/STD knowledge scale; score range 0-9; higher scores indicate greater HIV/STD knowledge
Self-efficacy | 12 months
  8-item self-efficacy for HIV prevention scale; score range 1-4; higher scores indicate greater self-efficacy
Condom Attitudes | 12 months
  3-item Condom Attitudes scale; score range 1-5; higher scores indicate greater condom attitudes
Condom Norms | 12 months
  3-item condom norms scale; score range 1-5; higher scores indicate greater condom norms
Communication intentions | 12 months
  1-item sexual communication intention; score range 0-4; higher scores indicate greater intentions to communicate with partners about sex
Condom use intention | 12 months
  1-item condom use intention; score range 0-4; higher scores indicate greater intentions to use condoms at next intercourse
sexual assertiveness | 12 months
  3-item sexual assertiveness scale score range 1-5; higher scores indicate greater sexual assertiveness

CONTACTS AND LOCATIONS:
Overall Officials: Laura Widman, PhD, Principal Investigator — North Carolina State University
Locations (1):
- North Carolina State University, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be available upon request with proper IRB training and approval
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available within 3 months of study completion.
Access Criteria: Contact the investigator: lmwidman@ncsu.edu